CLINICAL TRIAL: NCT06988345
Title: Outcome Juxtarenal Aortic Aneurysm After Open Repair
Brief Title: Juxtarenal Aortic Aneurysm
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: University Hospital Augsburg (Other); University Hospital, Aachen (Other); Goethe University (Other); University Hospital Heidelberg (Other); University Hospital Regensburg (Other); University of Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Univ.-Prof. Dr. med. Alexander Oberhuber, Univ.-Prof. Dr. med., University Hospital Muenster
Other Study IDs: 2023-641-f-S
Record Dates: First submitted 2024-11-20; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Juxtarenal Aneurysms; Open Repair

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
All patients with a juxtarenal abdominal aortic aneurysm who underwent open aneurysm therapy between January 2010 and July 2020 were included retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a juxtarenal aneurysm (defined as infrarenal neck <10mm and clamping above at least one renal artery [31592091])
* Open therapy with infrarenal (Anschluss)
* >18 years

Exclusion Criteria:

* Patients with an anastomosis above the renal arteries (e.g. including bypass to a renal artery)
* Patients with supravisceral clamping
* Patients with reconstruction of the aorta in the suprarenal area
* Patients with connective tissue diseases (e.g. Marfan syndrome or Ehler Danlos syndrome)
* Post-dissection aneurysms
* Infected aneurysms
* Conversions after endovascular therapy
* Inflammatory aneurysms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a juxtarenal aneurysm who fulfill the inclusion criteria or do not fulfill the exclusion criteria may be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days after intervention
  Mortality after 30 days postop
Acute renal failure | 30 days after intervention
  Acute renal failure postoperatively, defined by KDIGO criteria of AKI [22890468]

SECONDARY OUTCOMES:
Dialysis | during Follow up period, checked every year
  Permanent dialysis required
Reinterventions | during Follow up period, checked every year
  Rates of Reinterventions
Mortality | during Follow up period (up to 13 years)
  Overall mortality
Aneurysm-related Mortality | during Follow up period (up to 13 years)
  Aneurysm-related Mortality
Post-operative complication rates | During Follow-up period (up to 13 years)
  Post-operative complication rates:
  * cardiac
  * pulmonal
  * mesenterial
  * neurological
  * access-associated
  * re-intervention